CLINICAL TRIAL: NCT03893942
Title: Psychological Predictors of Post-surgical Recovery in Inflammatory Bowel Disease: a Pilot Cohort Study
Brief Title: Psychological Predictors in Colorectal IBD Surgery Recovery
Acronym: MIND-IBD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 2214
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Inflammatory Bowel Diseases; Mindfulness; Psychological predictors; Colorectal surgery
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone; Perceived Stress Scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires administration — Psychological and quality of life questionnaires
Other: Langer Mindfulness Scale (LMS) — The LMS is a 21-item questionnaire, assessing four domains associated with mindful thinking: novelty-seeking, engagement, novelty producing, and flexibility.
Other: Mindful Attention Awareness Scale (MAAS) — The MAAS is a 15-item questionnaire, designed to assess a core characteristic of dispositional mindfulness, namely, open or receptive awareness of and attention to what is taking place in the present
Other: Cognitive Flexibility Scale (CFS) — The CFS is 12-item self-report test assessing awareness.
Other: Life Orientation Test (LOT) — The LOT is a 10-item, self-administered scale assessing generalized expectancies for positive versus negative outcomes.
Other: Mini Locus of Control test (MLS) — The MLS is a 6-item questionnaire that includes 3 factors : chance, powerful others, and internality.
Other: Hospital Anxiety and Depression Scale (HADS) — The HADS is a 14-items rated on a four-point Likert scale. The questionnaire was designed to screen for the presence and severity of depression (HADS-D) and anxiety (HADS-A) in people with a physical symptomatology
Other: Perceived Stress Scale (PSS) — The PSS is 14-item self-report tool commonly used to provide a global measure of perceived stress in daily life.

SUMMARY:
This is an observation pilot trial aimed to study to the association between mindfulness and other psychological factors, including both protective and risk factors, with recovery of functional ability following colorectal surgery for Inflammatory Bowel Diseases (IBD), including Crohn's disease and Ulcerative Colitis.

DETAILED DESCRIPTION:
The chronic nature of Inflammatory Bowel Disease (IBD) leads to a significant impact on patients' lives, beyond intestinal symptoms alone. The sequelae of this can be seen in the increased rates of depression and reduced quality of life (QoL). Surgery may provide a way to effectively induce long-term symptoms remission, although there is a short postoperative transitory period whereas quality of life might decrease. Over the last years, increasing interest has been gained by perioperative recovery protocols, aiming to accelerate functional recovery and to reduce complications. Some of these protocols include an in-depth discussion with both dedicated nurses and/or surgeons to decrease surgery-associated stress reaction. Nevertheless, no one of the proposed protocols has included a psychological assessment in order to correlate it with functional recovery. We suggest that studying the psychological characteristics of the patients (with a specific focus on mindfulness) could lead to open a new research front to optimize patients' outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old (both males and females).
* Patients diagnosed with Inflammatory Bowel Disease (Crohn's Disease or Ulcerative Colitis).
* Patients scheduled for elective open or laparoscopic surgery for curative intent.

Exclusion Criteria:

* Patients unable to give the written informed consent.
* Patients < 18 years old.
* Patients undergoing surgery in emergency setting.
* Patients with pre-operative evidence of colorectal cancer or High Grade/Low grade dysplasia.
* Pregnant or breastfeeding patients.
* Any condition that, in the opinion of the investigator, can interfere with the study protocol (e.g. neuropsychiatric disorders or dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Inflammatory Bowel Disease (Crohn's Disease or Ulcerative Colitis) scheduled for elective curative colorectal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-04-16 (Actual); Primary Completion 2020-10-25 (Actual); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Correlation between psychological predictors questionnaires outcome and length of hospital stay | Post-operative day 7
  Length of stay calculated in days from the day of surgery until the day of discharge
Correlation between psychological predictors questionnaires outcome and quality of life | Post-operative day 30
  Quality of Life will be assessed by using the Short Inflammatory Bowel Disease Quality of Life Questionnaire (S_IBDQOL)
Correlation between psychological predictors questionnaires outcome and quality of life | Post-operative day 90
  Quality of Life will be assessed by using the Short Inflammatory Bowel Disease Quality of Life Questionnaire (S_IBDQOL)
Correlation between psychological predictors questionnaires outcome and quality of life | Post-operative month 6
  Quality of Life will be assessed by using the Short Inflammatory Bowel Disease Quality of Life Questionnaire (S_IBDQOL)
Correlation between psychological predictors questionnaires outcome and quality of life | Post-operative month 12
  Quality of Life will be assessed by using the Short Inflammatory Bowel Disease Quality of Life Questionnaire (S_IBDQOL)

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Spinelli, MD, PhD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- IRCCS Istituto Clinico Humanitas, Division of Colon and Rectal Surgery, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: No